CLINICAL TRIAL: NCT00748657
Title: A Phase II Trial of NCI-Supplied Agent: Bevacizumab (rhuMAB VEGF) (NSC# 704865) for Recurrent Sex Cord-Stromal Tumors of the Ovary
Brief Title: Bevacizumab in Treating Patients With Recurrent Sex Cord-Stromal Tumors of the Ovary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00611; NCI-2009-00611 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000613531; GOG-0251; GOG-0251 (Other: NRG Oncology); GOG-0251 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Malignant Ovarian Epithelial Tumor; Ovarian Granulosa Cell Tumor; Ovarian Gynandroblastoma; Ovarian Sertoli-Leydig Cell Tumor; Ovarian Sex Cord Tumor With Annular Tubules; Ovarian Sex Cord-Stromal Tumor; Ovarian Sex Cord-Stromal Tumor of Mixed or Unclassified Cell Types; Ovarian Steroid Cell Tumor
MeSH Terms: conditions — Granulosa cell tumor of the ovary; Ovarian gynandroblastoma; Sertoli-Leydig Cell Tumor | interventions — Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well bevacizumab works in treating patients with sex cord-stromal tumors of the ovary that have come back. Monoclonal antibodies, such as bevacizumab, may block tumor growth in different ways by targeting certain cells. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the anti-tumor activity of bevacizumab by assessing frequency of objective response in patients with recurrent sex cord-stromal tumors of the ovary who have measurable disease.

SECONDARY OBJECTIVES:

I. To determine the nature and degree of toxicity in these patients. II. To determine the overall survival and progression-free survival of these patients.

TERTIARY OBJECTIVES:

I. To quantify expression of angiogenic or lymphangiogenic markers in recurrent stromal tumors of the ovary to determine the frequency of alterations and potential utility of biologic agents directed at these proteins for inclusion in future studies.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with histologically confirmed recurrent ovarian stromal tumor (granulosa cell tumor, granulosa cell-theca cell tumor, Sertoli-Leydig cell tumor [androblastoma], steroid [lipid] cell tumor, gynandroblastoma, unclassified sex cord-stromal tumor, sex cord tumor with annular tubules)
* Patients must have measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) criteria

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each ?target? lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
* Patients must have a Gynecologic Oncology Group (GOG) performance grade of 0, 1, or 2
* Patients of childbearing potential must have a negative pregnancy test and must agree to practice an effective means of birth control
* Patients who have met the pre-entry requirements specified
* There are no restrictions on prior therapy; however, patients cannot have previously had treatment with bevacizumab
* Absolute neutrophil count (ANC) >= 1,000/?l
* Platelets greater than or equal to 75,000/?l
* Creatinine =< 1.5 x institutional upper limit normal (ULN)
* Bilirubin =< 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) less 2.5 x ULN
* Alkaline phosphatase less 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) version (v)3.0 grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) < 1.2 times the upper limit of normal
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with newly diagnosed disease
* Patients with serious non-healing wound, ulcer, or bone fracture
* Patients who have received prior therapy with bevacizumab or other inhibitors of vascular endothelial growth factor (VEGF)
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA), or subarachnoid hemorrhage within 6 months of the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
  * Myocardial infarction or unstable angina within 6 months prior to registration
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Serious cardiac arrhythmic requiring medication.
  * Grade 2 or greater peripheral vascular disease
* Patients with GOG performance grade of 3 or 4
* Patients with clinically significant peripheral arterial disease; e.g., claudication within 6 months
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients with clinically significant proteinuria; urine protein should be screened by urine protein-creatinine ratio (UPCR); the UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection; specifically; a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24 hour urine collection; obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24 hour urine); send sample to lab with request for urine protein and creatinine levels (separate requests); the lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL); the UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL); patients must have a UPCR < 1.0 to allow participation in the study
* Patients with a history of cardiovascular accident (CVA) within 6 months prior to registration
* Patients with any signs of bowel obstruction or patients who require parenteral hydration and/or nutrition
* Patients whose circumstances do not permit completion of the study or the required follow-up
* Patients who are pregnant or nursing; patients who may become pregnant must agree to use contraceptive measures during the study and for at least 3 months after the completion of bevacizumab therapy
* Patients who have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first date of treatment on this study, or anticipate the need for major surgical procedure during the course of the study; patients with placement of vascular access device or core biopsy within 7 days prior to the first date of treatment on this study
* Patients with active infection requiring parenteral antibiotics
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09-22 (Actual); Primary Completion 2013-01-31 (Actual); Study Completion 2013-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jubilee Brown, Principal Investigator — NRG Oncology
Locations (36):
- United States (36):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 9/22/2008 and closed to accrual on 1/31/2011 (suspended from 1/4/2010 to 8/9/2010).
Groups:
- Bevacizumab: Bevacizumab 15 mg/kg IV every 21 days until disease progression or adverse effects prohibit further treatment
Period: Overall Study
Arm/Group | Bevacizumab
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligibile and treatmed patients
Arm/Group | Bevacizumab
Number analyzed (Participants) | 36
Age, Customized [Number; unit: participants]
  20-29 | 0
  30-39 | 1
  40-49 | 8
  50-59 | 12
  60-69 | 11
  70-79 | 4
  80-89 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.0
Time Frame: Every other cycle for 6 months; then every 3 months for two years; then every six months for three years; and at any other time if clinically indicated based on symptoms, physical signs suggestive of progressive disease or rising serum tumor maker levels
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Bevacizumab
Number analyzed (Participants) | 36
percentage of patients | 16.7 [7.5 to 30.3]

2. Secondary Outcome: Progression-free Survival
Description: Progression-Free Survival is the period from study entry until disease progression, death or date of last contact.
Time Frame: as for outcome 1
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 36
Months | 9.3 [4.1 to 15.0]

3. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 36
Months | NA [44.9 to NA] — NA (not available): median OS was not reached but is >65.9 months, as is the upper bound of the 95% CI.

4. Secondary Outcome: Number of Participants With Episodes and Grade of Adverse Events as Assessed by Common Terminology for Adverse Events Version 3.0
Description: Adverse Events at least possibly related to study agent.
Time Frame: Up to 5 years
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE (adverse event).
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36
Participants
  Leukopenia | 32 | 2 | 1 | 1 | 0 | 0
  Thrombocytopenia | 28 | 8 | 0 | 0 | 0 | 0
  Anemia | 21 | 7 | 7 | 1 | 0 | 0
  Other Hematologic | 33 | 2 | 1 | 0 | 0 | 0
  Allergy/Immunology | 23 | 11 | 2 | 0 | 0 | 0
  Auditory/Ear | 29 | 0 | 6 | 1 | 0 | 0
  Cardiac | 15 | 6 | 9 | 5 | 1 | 0
  Coagulation | 35 | 0 | 0 | 1 | 0 | 0
  Constitutional | 12 | 10 | 13 | 1 | 0 | 0
  Dermatologic | 17 | 14 | 4 | 1 | 0 | 0
  Endocrine | 33 | 2 | 1 | 0 | 0 | 0
  Gastrointestinal | 6 | 10 | 15 | 5 | 0 | 0
  Genitourinary/Renal | 29 | 5 | 1 | 1 | 0 | 0
  Hemorrhage | 17 | 18 | 0 | 1 | 0 | 0
  Infection | 23 | 0 | 11 | 2 | 0 | 0
  Lymphatics | 31 | 4 | 1 | 0 | 0 | 0
  Metabolic | 13 | 10 | 8 | 3 | 2 | 0
  Musculoskeletal | 30 | 5 | 1 | 0 | 0 | 0
  Neurosensory | 21 | 13 | 1 | 1 | 0 | 0
  Other Neurological | 22 | 12 | 1 | 1 | 0 | 0
  Ocular/Visual | 30 | 6 | 0 | 0 | 0 | 0
  Pain | 1 | 11 | 16 | 8 | 0 | 0
  Pulmonary | 12 | 20 | 1 | 3 | 0 | 0
  Sexual/Reproductive | 32 | 4 | 0 | 0 | 0 | 0
  Syndromes | 35 | 1 | 0 | 0 | 0 | 0
  Vascular | 35 | 0 | 1 | 0 | 0 | 0
  Death, Not CTC coded | 35 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 13/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=36)
Tinnitus (Ear and labyrinth disorders) | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Ulcer,gi - Stomach (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Syncope (Nervous system disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 1
Pain: Tumor (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=36)
Allergy/Immunology - Other (Immune system disorders) | 1
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Rhinitis (Immune system disorders) | 11
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 6
Platelets (Blood and lymphatic system disorders) | 8
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 15
Palpitations (Cardiac disorders) | 4
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 16
Pericardial Effusion (Cardiac disorders) | 1
Inr (Vascular disorders) | 1
Constitutional Symptoms - Other (General disorders) | 2
Sweating (General disorders) | 1
Weight Gain (General disorders) | 1
Fever (General disorders) | 3
Weight Loss (General disorders) | 5
Rigors/Chills (General disorders) | 3
Fatigue (General disorders) | 23
Insomnia (General disorders) | 3
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 2
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 5
Bruising (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 12
Dry Skin (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3
Flushing (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Hot Flashes (Endocrine disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Heartburn (Gastrointestinal disorders) | 3
Ulcer,gi - Stomach (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 3
Taste Alteration (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 4
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 10
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 22
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 13
Hemorrhage, Gu - Vagina (Vascular disorders) | 1
Hemorrhage/Pulmonary - Bronchopulmonary Nos (Vascular disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 2
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 15
Hematoma (Vascular disorders) | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 2
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Ureter (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Edema: Limb (Blood and lymphatic system disorders) | 5
Ast (Metabolism and nutrition disorders) | 7
Gfr (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 4
Cholesterol,serum High (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 6
Creatinine (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Ggt (Metabolism and nutrition disorders) | 2
Alt (Metabolism and nutrition disorders) | 4
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5
Bilirubin (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Trismus (Musculoskeletal and connective tissue disorders) | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 5
Mood Alteration - Anxiety (Nervous system disorders) | 7
Mood Alteration - Agitation (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Neuropathy-Sensory (Nervous system disorders) | 15
Watery Eye (Eye disorders) | 1
Dry Eye (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Blurred Vision (Eye disorders) | 4
Pain - Other (General disorders) | 3
Pain: Urethra (General disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Vagina (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 3
Pain: Chest Wall (General disorders) | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 1
Pain: Head/Headache (General disorders) | 23
Pain: Neck (General disorders) | 4
Pain: Extremity-Limb (General disorders) | 7
Pain: Back (General disorders) | 7
Pain: Joint (General disorders) | 9
Pain: Kidney (General disorders) | 1
Pain: Bladder (General disorders) | 1
Pain: Pain Nos (General disorders) | 1
Pain: Stomach (General disorders) | 1
Pain: Oral Cavity (General disorders) | 4
Pain: Abdominal Pain Nos (General disorders) | 18
Pain: Oral - Gums (General disorders) | 2
Pain: Skin (General disorders) | 1
Pain: Middle Ear (General disorders) | 1
Pain: Face (General disorders) | 1
Pain: Tumor (General disorders) | 1
Pain: Liver (General disorders) | 1
Pain: Muscle (General disorders) | 3
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 3
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 7
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Cystitis (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 5
Libido (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 2
Flu-Like Syndrome (General disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less